CLINICAL TRIAL: NCT01075984
Title: Pharmacokinetics, Safety, and Tolerability of Intravenous Posaconazole Solution Followed by Oral Posaconazole Suspension (SCH 56592) in Subjects at High Risk for Invasive Fungal Infections (Phase 1b; Protocol No. P05520)
Brief Title: Pharmacokinetics, Safety, and Tolerability of Intravenous Posaconazole Solution Followed by Oral Posaconazole Suspension in Subjects at High Risk for Invasive Fungal Infections (P05520)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P05520
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Fungal Infection
Keywords: Antifungal Agents pharmacokinetics; Mycoses prevention and control
MeSH Terms: conditions — Mycoses | interventions — posaconazole; Glucose; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- POS IV 200 mg single dose (Cohort 0) (Active Comparator): POS 200 mg IV single dose infused over 1.5 hours on Day 1 followed 12 hours later by POS oral 400 mg, then by POS oral 400 mg BID on Days 2 through 6 and a single morning dose on Day 7 (Cohort 0)
  Interventions: Drug: Posaconazole
- Dextrose 5% in water (Cohort 0) (Placebo Comparator): Placebo IV single dose infused over 1.5 hours on Day 1 followed 12 hours later by POS oral 400 mg, then by POS oral 400 mg BID on Days 2 through 6 and a single morning dose on Day 7 (Cohort 0)
  Interventions: Drug: Posaconazole; Drug: Dextrose 5% in water
- POS IV 200 mg BID (Cohort 1) (Experimental): POS 200 mg IV infused over 1.5 hours BID on Day 1, followed by POS 200 mg IV once daily on Days 2 through 14, then by POS 400 mg oral BID through Day 28 (Cohort 1)
  Interventions: Drug: Posaconazole
- POS IV 300 mg BID (Cohort 2) (Experimental): POS 300 mg IV infused over 1.5 hours BID on Day 1, followed by POS 300 mg IV once daily on Days 2 through 14, then by POS 400 mg oral BID through Day 28 (Cohort 2). After Day 5, POS IV was administered continuously or intermittently, depending on oral tolerability.
  Interventions: Drug: Posaconazole
- POS IV 300 mg BID (Cohort 3) (Experimental): POS 300 mg IV infused over 1.5 hours BID on Day 1, followed by POS 300 mg IV once daily on Days 2 through 5, then by POS 200 mg oral TID or POS 400 mg oral BID through Day 28, or POS 200-300 mg IV once daily as required (Cohort 3). After Day 5, POS IV was administered continuously or intermittently, depending on oral tolerability.
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole
  Other Names: SCH 056592
Drug: Dextrose 5% in water
  Other Names: SCH 056592 (2)
  Arms: Dextrose 5% in water (Cohort 0)

SUMMARY:
The purpose of this study is to collect pharmacokinetic (PK) information related to how well intravenous Posaconazole (POS IV), is distributed in the body and to determine the safety and tolerability of this new formulation. In addition, the PK, safety, and tolerability of switching from taking POS IV to taking Posaconazole Oral Suspension (POS Oral) will be evaluated. The data collected in this study will be compared to data collected in previous studies.

Individuals who have been diagnosed by their physicians with a blood disease or cancer that can affect their infection-fighting white blood cells will be asked to participate in the trial. Since these blood diseases and their treatments can weaken the immune system, they may put these individuals at a high risk for getting a serious fungal infection of their internal organs or blood (invasive fungal infection). As these fungal infections can be hard to detect early and can be life-threatening, many physicians believe that individuals diagnosed with these diseases should receive antifungal therapy to try to lower their risk of getting this type of infection.

Enrollment into this study will take place in several stages (cohorts). The determination of which cohort an individual will be asked to participate in is based on which cohort is open at the site at the time the individual is approached to consider study participation.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects greater than or equal to 18 years of age (weighing greater than 34 kg [75 lb]), of either sex and of any race/ethnicity.
* Disease definition for each subject: Anticipated (likely to develop within 3 days to 5 days) or documented prolonged neutropenia (absolute neutrophil count [ANC] <500/mm^3 [0.5 x 10^9/L]) at Baseline and likely to last for at least 7 days due to:

  * a. Standard intensive chemotherapy, anthracycline-based or other accepted regimen (excluding any investigational agent), for a new diagnosis of acute myelogenous leukemia (AML);
  * b. Chemotherapy for AML in first relapse; or
  * c. Therapy for myelodysplastic syndromes in transformation to AML or other diagnoses of secondary AML (therapy related, antecedent hematological disorders) or chronic myelogenous leukemia in blast crisis
* Disease definition for each Cohort 3 subject: In addition to subjects defined above, allogeneic hematopoietic stem cell transplant (HSCT) subjects may be randomized in either the pre-engraftment period (i.e., after they have received their conditioning regimen for the transplant, but while they are still neutropenic) or in the post-engraftment period if they are receiving immunosuppressive therapy for prevention or treatment of graft-versus-host disease (e.g., steroids, tacrolimus, cyclosporin, mycophenolate mofetil, and antithymocyte globulin).

Exclusion Criteria:

* A female subject must not be pregnant, must not intend to become pregnant during the study, or must not be nursing.
* Excluded prior treatments. A subject must not have received systemic antifungal therapy (oral, intravenous, or inhaled) for the treatment of proven or probable IFI within 30 days of Enrollment.
* A subject must not have moderate or severe liver dysfunction at Baseline, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels greater than three times the upper limit of normal (ULN), AND a total bilirubin level greater than two times the ULN. For Cohorts 1 and 2, a subject must not have a known or suspected history of Gilbert's disease.
* A subject must not have an electrocardiogram (ECG) with a prolonged QTc interval by manual reading: QTc greater than 500 msec.
* A subject must not have prior enrollment in this study, or other POS studies within 90 days of study entry.
* A subject must not have a known or suspected invasive or systemic fungal infection at Baseline. Those subjects receiving empiric anti-fungal therapy within 7 days prior to Baseline must have had a diagnostic work-up that ruled out a possible invasive fungal infection.
* A subject must not have creatinine clearance levels (measured or calculated) below 50 mL/min.
* A subject must not have a history of Type I hypersensitivity or idiosyncratic reactions to azole agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2010-02-23 (Actual); Primary Completion 2012-11-20 (Actual); Study Completion 2012-11-20 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Maertens J, Cornely OA, Ullmann AJ, Heinz WJ, Krishna G, Patino H, Caceres M, Kartsonis N, Waskin H, Robertson MN. Phase 1B study of the pharmacokinetics and safety of posaconazole intravenous solution in patients at risk for invasive fungal disease. Antimicrob Agents Chemother. 2014 Jul;58(7):3610-7. doi: 10.1128/AAC.02686-13. Epub 2014 Apr 14. PMID 24733463
- [Result] Cornely OA, Robertson MN, Haider S, Grigg A, Geddes M, Aoun M, Heinz WJ, Raad I, Schanz U, Meyer RG, Hammond SP, Mullane KM, Ostermann H, Ullmann AJ, Zimmerli S, Van Iersel MLPS, Hepler DA, Waskin H, Kartsonis NA, Maertens J. Pharmacokinetics and safety results from the Phase 3 randomized, open-label, study of intravenous posaconazole in patients at risk of invasive fungal disease. J Antimicrob Chemother. 2017 Dec 1;72(12):3406-3413. doi: 10.1093/jac/dkx263. PMID 28961714

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who started the study were eligible to enter the follow-up phase, whether or not they completed the treatment phase.
Groups:
- Posaconazole (POS) 200 mg IV Single Dose (Cohort 0): POS 200 mg IV single dose on Day 1 followed 12 hours later by POS oral 400 mg, then by POS oral 400 mg BID on Days 2 through 6 and a single morning dose on Day 7 (Cohort 0)
- Placebo IV Single Dose (Cohort 0): Placebo IV single dose on Day 1, followed 12 hours later by POS oral 400 mg, then by POS oral 400 mg BID on Days 2 through 6 and a single morning dose on Day 7 (Cohort 0)
- POS 200 mg IV BID (Cohort 1): POS 200 mg IV BID on Day 1, followed by POS 200 mg IV once daily on Days 2 through 14, then by POS 400 mg oral BID through Day 28 (Cohort 1)
- POS 300 mg IV BID (Cohort 2): POS 300 mg IV BID on Day 1, followed by POS 300 mg IV once daily on Days 2 through 14, then by POS 400 mg oral BID through Day 28 (Cohort 2). After Day 5, POS IV was administered continuously or intermittently, depending on oral tolerability.
- POS 300 mg IV BID (Cohort 3): POS 300 mg IV BID on Day 1 followed by POS 300 mg IV once daily on Days 2 through 5, then by POS 200 mg oral TID or POS 400 mg oral BID through Day 28 or POS 200-300 mg IV once daily as required (Cohort 3). After Day 5, POS IV was administered continuously or intermittently, depending on oral tolerability.
Period: Treatment Phase
Arm/Group | Posaconazole (POS) 200 mg IV Single Dose (Cohort 0) | Placebo IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2) | POS 300 mg IV BID (Cohort 3)
Started | 10 | 11 | 21 | 24 | 213
Completed | 10 | 10 | 14 | 17 | 153
Not Completed | 0 | 1 | 7 | 7 | 60
Not completed — Adverse Event | 0 | 1 | 3 | 7 | 35
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 15
Not completed — Treatment Failure | 0 | 0 | 1 | 0 | 5
Not completed — Progression of disease | 0 | 0 | 0 | 0 | 2
Period: Follow-up Phase
Arm/Group | Posaconazole (POS) 200 mg IV Single Dose (Cohort 0) | Placebo IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2) | POS 300 mg IV BID (Cohort 3)
Started | 10 | 10 | 20 (One participant did not start the follow-up phase for reasons unrelated to study procedures.) | 21 (Three participants did not start the follow-up phase: one died and two were lost to follow-up.) | 212 (One participant withdrew consent before the start of the follow-up phase.)
Completed | 10 | 10 | 19 | 19 | 165
Not Completed | 0 | 0 | 1 | 2 | 47
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 27
Not completed — Administrative | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 10
Not completed — Progression of disease | 0 | 0 | 0 | 0 | 2
Not completed — Treatment failure | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- POS 200 mg IV Single Dose (Cohort 0): POS 200 mg IV single dose on Day 1 followed 12 hours later by POS oral 400 mg, then by POS oral 400 mg BID on Days 2 through 6 and a single morning dose on Day 7 (Cohort 0)
- Total: Total of all reporting groups
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | Placebo IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2) | POS 300 mg IV BID (Cohort 3) | Total
Number analyzed (Participants) | 10 | 11 | 21 | 24 | 213 | 279
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (17.4) | 59.5 (12.3) | 49.1 (14.7) | 52.4 (13.4) | 50.7 (14.7) | 51.3 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 8 | 11 | 96 | 126
  Male | 5 | 5 | 13 | 13 | 117 | 153

OUTCOME MEASURES:

1. Primary Outcome: Single Dose Trough Concentration of IV Posaconazole (Cmin)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: 12 hours after start of infusion on Day 1 (Cohorts 0, 1 and 2)
Population: The PK-evaluable population included participants who had no major protocol violations and had documented adherence to the dosing and PK regimens. Cohort 3 was not evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2)
Number analyzed (Participants) | 10 | 20 | 22
ng/mL | 318 (107) | 295 (113) | 467 (172)

2. Primary Outcome: Steady State Trough Concentration of IV Posaconazole (Cmin)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: 24 hours after start of infusion on Day 14 (Cohorts 1 and 2), or Day 10 (Cohort 3)
Population: The PK-evaluable population included participants who had no major protocol violations and had documented adherence to the dosing and PK regimens.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2) | POS 300 mg IV BID (Cohort 3)
Number analyzed (Participants) | 15 | 19 | 30
ng/mL | 958 (605) | 1046 (515) | 1164 (462)

3. Primary Outcome: Single Dose Maximum Concentration of IV Posaconazole (Cmax)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: Predose and 1, 1.5, 1.75, 4, 8, and 12 hours after start of infusion on Day 1 (Cohorts 0, 1 and 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2)
Number analyzed (Participants) | 10 | 20 | 22
ng/mL | 881 (334) | 990 (467) | 1590 (980)

4. Primary Outcome: Steady State Maximum Concentration of IV Posaconazole (Cmax)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: Predose and 1, 1.5, 1.75, 4, 8, and 12 hours after start of infusion on Day 14 (Cohorts 1 and 2), or Day 10 (Cohort 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2) | POS 300 mg IV BID (Cohort 3)
Number analyzed (Participants) | 15 | 19 | 30
ng/mL | 1947 (966) | 2610 (1010) | 3696 (2950)

5. Primary Outcome: Single Dose Time of Observed Maximum Concentration of IV Posaconazole (Tmax)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: Predose and 1, 1.5, 1.75, 4, 8, and 12 hours after start of infusion on Day 1 (Cohorts 0 and 1)
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2)
Number analyzed (Participants) | 10 | 20 | 22
Hours | 1.42 [0.95 to 1.78] | 1.48 (50) [1.00 to 3.97] | 1.54 [1.00 to 1.92]

6. Primary Outcome: Steady State Time of Observed Maximum Concentration of IV Posaconazole (Tmax)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: Predose and 1, 1.5, 1.75, 4, 8, and 12 hours after start of infusion on Day 14 (Cohorts 1 and 2), or Day 10 (Cohort 3)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2) | POS 300 mg IV BID (Cohort 3)
Number analyzed (Participants) | 15 | 19 | 30
Hours | 1.00 (50) [1.00 to 4.02] | 1.50 (39) [0.98 to 4.00] | 1.52 (80) [1.00 to 2.00]

7. Primary Outcome: Single Dose Area Under the Concentration Versus Time Curve of IV Posaconazole (AUC)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: Predose and 1, 1.5, 1.75, 4, 8, and 12 hours after start of infusion on Day 1 (Cohorts 0, 1 and 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2)
Number analyzed (Participants) | 10 | 20 | 22
hour*ng/mL | 5940 (2190) | 5390 (1540) | 8240 (2140)

8. Primary Outcome: Steady State Area Under the Concentration Versus Time Curve of IV Posaconazole (AUC)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: Predose and 1, 1.5, 1.75, 4, 8, 12, and 24 hours after start of infusion on Day 14 (Cohorts 1 and 2), or Day 10 (Cohort 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2) | POS 300 mg IV BID (Cohort 3)
Number analyzed (Participants) | 15 | 19 | 30
hour*ng/mL | 28241 (14511) | 33754 (14196) | 37586 (11504)

9. Primary Outcome: Steady State Average Concentration of IV Posaconazole (Cavg)
Description: Blood samples were collected from participants for the determination of plasma POS concentration. Cavg was calculated as steady state AUC / dosing interval (24 hours).
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2) | POS 300 mg IV BID (Cohort 3)
Number analyzed (Participants) | 15 | 19 | 30
ng/mL | 1180 (605) | 1410 (592) | 1566 (479)

10. Primary Outcome: Steady State Total Body Clearance of IV Posaconazole (CL)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: Predose and 1, 1.5, 1.75, 4, 8, and 12 hours after start of infusion on Day 14 (Cohorts 1 and 2), or Day 10 (Cohort 3)
Population: CL for posaconazole was not calculated in this study because it was collected in other studies more appropriate for evaluation of this parameter.
Arm/Group | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2) | POS 300 mg IV BID (Cohort 3)
Number analyzed (Participants) | 0 | 0 | 0

11. Primary Outcome: Steady State Trough Concentration of Oral Posaconazole (Cmin)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: 12 hours after dosing on Day 7 (Cohort 0), or Day 28 (Cohorts 1 and 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2)
Number analyzed (Participants) | 15 | 7 | 4
ng/mL | 370 (125) | 532 (266) | 316 (164)

12. Primary Outcome: Steady State Maximum Concentration of Oral Posaconazole (Cmax)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: Predose and 3, 5, 8 and 12 hours after dosing on Day 7 (Cohort 0), or Day 28 (Cohorts 1 and 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2)
Number analyzed (Participants) | 15 | 7 | 4
ng/mL | 494 (176) | 811 (208) | 430 (260)

13. Primary Outcome: Steady State Time of Observed Maximum Concentration of Oral Posaconazole (Tmax)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: Predose and 3, 5, 8 and 12 hours after dosing on Day 7 (Cohort 0), or Day 28 (Cohorts 1 and 2)
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2)
Number analyzed (Participants) | 15 | 7 | 4
Hours | 3.03 [2.73 to 5.13] | 3.05 (50) [0 to 8.13] | 5.54 (39) [2.97 to 11.62]

14. Primary Outcome: Steady State Area Under the Concentration Versus Time Curve of Oral Posaconazole (AUC)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: Predose and 3, 5, 8 and 12 hours after dosing on Day 7 (Cohort 0), or Day 28 (Cohorts 1 and 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2)
Number analyzed (Participants) | 15 | 7 | 4
hour*ng/mL | 5080 (1700) | 6920 (1910) | 3970 (2050)

15. Primary Outcome: Steady State Average Concentration of Oral Posaconazole (Cavg)
Description: Blood samples were collected from participants for the determination of plasma POS concentration. Cavg was calculated as steady state AUC / dosing interval (12 hours).
Time Frame: Predose and 3, 5, 8 and 12 hours after dosing on Day 7 (Cohort 0), or Day 28 (Cohorts 1 and 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2)
Number analyzed (Participants) | 15 | 7 | 4
ng/mL | 423 (144) | 570 (160) | 331 (172)

16. Primary Outcome: Steady State Apparent Total Body Clearance of Oral Posaconazole (CL/F)
Description: Blood samples were collected from participants for the determination of plasma POS concentration.
Time Frame: Predose and 3, 5, 8 and 12 hours after dosing on Day 7 (Cohort 0), or Day 28 (Cohorts 1 and 2)
Population: CL/F for posaconazole was not calculated in this study because it was collected in other studies more appropriate for evaluation of this parameter
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 14 (Cohort 0); Up to Day 35 (Cohorts 1, 2, and 3)
Groups:
- POS 300 mg IV BID (Cohort 2 and 3): POS 300 mg IV BID on Day 1, followed by POS 300 mg IV once daily on Days 2 through 14, then by POS 400 mg oral BID through Day 28 (Cohort 2); POS 300 mg IV BID on Day 1 followed by POS 300 mg IV once daily on Days 2 through 5, then by POS 200 mg oral TID or POS 400 mg oral BID through Day 28 or POS 200-300 mg IV once daily as required (Cohort 3). After Day 5, POS IV was administered continuously or intermittently, depending on oral tolerability.
Arm/Group | POS 200 mg IV Single Dose (Cohort 0) | Placebo IV Single Dose (Cohort 0) | POS 200 mg IV BID (Cohort 1) | POS 300 mg IV BID (Cohort 2 and 3)
Serious Adverse Events (participants affected / at risk) | 2/10 | 2/11 | 4/21 | 71/237
Other Adverse Events (participants affected / at risk) | 10/10 | 11/11 | 20/21 | 229/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POS 200 mg IV Single Dose (Cohort 0) (N=10) | Placebo IV Single Dose (Cohort 0) (N=11) | POS 200 mg IV BID (Cohort 1) (N=21) | POS 300 mg IV BID (Cohort 2 and 3) (N=237)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Graft versus host disease in intestine (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Graft versus host disease in lung (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningoencephalitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Smear cervix abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelitis transverse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Venoocclusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POS 200 mg IV Single Dose (Cohort 0) (N=10) | Placebo IV Single Dose (Cohort 0) (N=11) | POS 200 mg IV BID (Cohort 1) (N=21) | POS 300 mg IV BID (Cohort 2 and 3) (N=237)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 22 (39)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (9) | 5 (6) | 6 (8) | 52 (66)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 24 (51)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 17 (18)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 15 (18)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 14 (14)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 41 (46)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (4) | 25 (25)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 30 (36)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (5) | 6 (18) | 92 (131)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 17 (17)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 5 (5)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 6 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 7 (8)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 10 (10)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 13 (13)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 9 (11)
Nausea (Gastrointestinal disorders) | 2 (3) | 5 (5) | 9 (10) | 67 (77)
Oedema mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 15 (15)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (7)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (4) | 5 (6) | 2 (2) | 42 (48)
Catheter site erythema (General disorders) | 0 (0) | 1 (2) | 2 (3) | 15 (18)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 14 (15)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 38 (47)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 24 (25)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0) | 2 (2) | 44 (47)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 15 (16)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 0 (0) | 35 (39)
Pyrexia (General disorders) | 0 (0) | 3 (4) | 6 (6) | 69 (96)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 7 (7)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 6 (7)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 7 (7)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 14 (14)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Puncture site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 9 (10)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 13 (13)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 6 (6)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 14 (14)
Antithrombin III decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 12 (12)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 29 (32)
Fluid retention (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 7 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 2 (2) | 12 (12)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 5 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 8 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 3 (4) | 67 (77)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 30 (34)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (5) | 21 (24)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 17 (17)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 19 (21)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 10 (10)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 16 (20)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 14 (14)
Headache (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2) | 49 (53)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (3) | 56 (71)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (3) | 2 (4) | 12 (15)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 26 (29)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 14 (16)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 13 (14)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 7 (8)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 17 (18)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (6) | 31 (32)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 23 (26)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 2 (2) | 40 (52)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 17 (18)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 13 (18)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 24 (26)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts.